CLINICAL TRIAL: NCT06357403
Title: Association of Anti-factor Xa Activity With Venous Thromboembolism in Critically Ill Patients: a Prospective Multicentre Cohort Study
Brief Title: Association of Anti-factor Xa Activity With Venous Thromboembolism in Critically Ill Patients
Acronym: AntiXa-ICU
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva Schaden, Assoc. Prof. Dr., Medical University of Vienna
Other Study IDs: AntiXa-ICU 1881/2023
Record Dates: First submitted 2024-02-19; First posted 2024-04-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Thrombosis; Pulmonary Embolism; Enoxaparin
MeSH Terms: conditions — Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intensive care unit patients: Patients who are admitted to an participating intensive care unit who do not receive therapeutic anticoagulation.
  Interventions: Diagnostic Test: Anti-factor Xa activity calibrated for enoxaparin

INTERVENTIONS:
Diagnostic Test: Anti-factor Xa activity calibrated for enoxaparin — Anti-factor Xa activity calibrated for enoxaparin

SUMMARY:
The goal of this observational study is to analyse the association between anti-factor Xa activity (antiXa) and the occurence of venous thromboembolism (VTE; either deep vein thrombosis and/or pulmonary embolism) in critically ill patients who are admitted to an intensive care unit. The main questions it aims to answer are:

* What is the association between antiXa and VTE?
* What is the association between antiXa and symptomatic, respectively incidental, VTE?
* How is pharmacological anticoagulation with enoxaparin related to measured antiXa?
* What is the association between antiXa and bleeding complications.
* What is the incidence of venous thromboembolism in patients treated at an intensive care unit?
* How is the occurence of VTE related to patient-centred outcomes such as mortality, quality of life, length of stay and days outside of the intensive care unit/hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years at the time of intensive care unit admission
* Admission to a participating intensive care unit within the last 24 hours
* Expected discharge is later than 48 hours after enrolment

Exclusion Criteria:

* Therapeutic anticoagulation, defined as enoxaparin dose of at least 100 IE/kg when given twice daily or of at least 150 IE/kg when given once daily
* Extracorporeal membrane oxygenation in place or planned within 48 hours of study enrolment
* Planned regular administration of vitamin K antagonists, unfractionated heparin, low molecular weight heparin other than enoxaparin, thrombin inhibitors or factor X inhibitors within the observation period
* Estimated life expectancy below 48 hours or comfort terminal care order in place
* Previously diagnosed heparin-induced thrombocytopenia
* Pre-operative admission for elective surgery
* Previous enrolment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to an surgical or medical intensive care unit who do not receive therapeutic anticoagulation
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with new-onset venous thromboembolism | until discharge from the intensive care unit or up to 14 days after study inclusion
  New-onset deep vein thrombosis and/or new-onset pulmonary embolism. Both symptomatic and incidental events are included.

SECONDARY OUTCOMES:
Number of patients with new-onset upper extremity deep vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset lower extremity deep vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset central vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset symptomatic upper extremity deep vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset symptomatic lower extremity deep vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset incidental upper extremity deep vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset incidental lower extremity deep vein thrombosis | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset pulmonary embolism | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset symptomatic pulmonary embolism | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with new-onset incidental pulmonary embolism | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of patients with venous thromboembolism | prevalent at study enrolment
Number of patients with deep vein thrombosis | prevalent at study enrolment
Number of patients with pulmonary embolism | prevalent at study enrolment
Number of patients with new-onset venous thromboembolism | 90 days after study enrolment
Number of days with any bleeding | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of days with major and/or fatal bleeding | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of red blood cell concentrates administered | until discharge from the intensive care unit or up to 14 days after study inclusion
Number of days on which either procoagulant medication, platelet transfusion or fresh frozen plasma was administered | until discharge from the intensive care unit or up to 14 days after study inclusion
Length of stay in the intensive care unit | 90 days after study enrolment
Length of stay in the hospital | 90 days after study enrolment
Death | 90 days after study enrolment
Days alive and out of the intensive care unit | 90 days after study enrolment
Days alive and out of the hospital | 90 days after study enrolment
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) index value | 90 days after study enrolment
  Minimum -1.0, Maximum 1.0; An index value of 1.0 indicates the best possible state of health. Index values below 0.0 indicate the worst possible state of health.
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) visual analogue scale | 90 days after study enrolment
  Minimum 0. Maximum 100. A value of 0 indicates the worst possible state of health while a value of 100 indicates the best possible state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Schaden, MD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Department of Internal Medicine, Medical University of Graz, Graz, Styria
  - Department of Anaesthesia, Intensive Care Medicine and Pain Medicine, Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Undecided